CLINICAL TRIAL: NCT03490877
Title: Quantification of Scratch and Sleep in Atopic Dermatitis
Brief Title: Scratch and Sleep Quantification in Atopic Dermatitis
Acronym: SQUAD
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Lisa Beck, Professor, University of Rochester
Other Study IDs: SQUAD1.0
Record Dates: First submitted 2018-03-20; First posted 2018-04-06 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Atopic Dermatitis; Pruritus; Sleep Disturbance
Keywords: Atopic Dermatitis; Pruritus; Sleep Disturbance
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Parasomnias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atopic dermatitis (AD) is a chronic type of eczema affecting approximately 10% of adults and 12% of children in the US. The intense itching (pruritus) associated with AD can be significantly disruptive to sleep and quality of life for both the patients and their caregivers. AD is challenging to describe and measure. The purpose of this study is to see if we can reliably measure how much people with AD scratch and how scratching interferes with sleep and quality of life by using digital sensors, sleep studies and patient-reported information.

DETAILED DESCRIPTION:
Wrist worn accelerometers, sleep sensors, polysomnography (PSG), and associated data analysis platforms would provide quantitative and qualitative knowledge regarding the action of scratching and sleep quantity in a symptomatic atopic dermatitis (AD) population. Our overall aim is to validate the use of accelerometry technology and digital measures to quantitatively and qualitatively evaluate scratch and sleep in AD patients in a home environment.

Accelerometry devices appear similar to a wristwatch. The subject will be asked to wear an accelerometry device on each wrist during the study. The accelerometry device provides continuous measures of wrist activity and will be used to quantify nocturnal scratching and sleep behaviors to be compared to videography (annotated for scratch), sleep sensor, PSG and traditional patient-reported outcome (PRO) and Quality of Life (QoL) measures [Peak Pruritus Numerical Scale, Severity of Pruritus Scale (SPS), Patient Global Impression of Severity (PGIS), Medical Outcomes Study (MOS) Sleep Scale, Itch and Sleep Diary, Patient-Oriented Eczema Measure (POE), Patient-Reported Outcomes Measurement Information System (PROMIS)-pain interference, PROMIS- anxiety, Dermatology Life Quality Index (DLQI), Family Dermatology Life Quality Index (FDLQI), Children's Dermatology Life Quality Index (CDLQI), Device and Device Comfort Questionnaire] in patients with AD in a clinic and home setting in a well-controlled clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged > 12 to 75 years of age at the screening visit.
* Written informed consent from participant (and parent/guardian for those subjects under 18 years of age) and able to understand and cooperate with study instructions, visits and procedures.
* Native English speakers or fluent in English (per investigator's judgment)
* Has a clinical diagnosis of AD according to the criteria of Hanifin and Rajka (concomitant atopic dermatitis treatments are permitted on study).
* Has AD involvement ≥ 5% Body Surface Area (BSA), excluding the scalp.
* Has an Investigator's Static Global Assessment (ISGA) score of Mild (2), Moderate (3), or Severe (4) at the Screening Visit
* Have a minimum Peak Pruritus Numerical Rating Score (NRS) of 3 and/or Severity of Pruritus Scale (SPS) score of 1.
* Willingness to abstain from alcohol and illicit drugs on the day of the second overnight in-clinic study visit.

Exclusion Criteria:

* Has any clinically significant medical disorder, condition, disease or clinically significant physical examination finding at screening that in the Investigator's or designee's opinion may interfere with study objectives (e.g., expose subject to unacceptable risk by study participation, confound evaluation, result in adverse events, or interfere with subject's ability to complete the study).
* Has documented sleep apnea and/or other sleep related disorders (e.g., narcolepsy, restless legs syndrome, circadian rhythm disorder) or has a Body Mass Index (BMI) >35.
* Subject scores <15 on the Asthma Control Test (ACT; Appendix C), indicating poorly controlled asthma.
* Current shift worker or travel across more than two time zones in the past 2 weeks. (NOTE: for this travel criterion, subjects may enroll in the study if they delay enrollment until two weeks has lapsed since their travel).
* If the patient has significant eczema at the location where the bilateral wrist devices will need to be worn, making the devices intolerable for the patient, and in the opinion of the patient or investigator would likely lead to noncompliance.
* Has a significant active systemic or localized infection, including actively infected AD.
* If subject has a history of angioedema or anaphylaxis, has not had any anaphylactic reactions within the past 6 months.
* Has recently (within 30 days of the Screening Visit) participated in or is currently involved in another drug or device research study.
* Has any planned surgical or medical procedure that would overlap with study participation.
* Is a female who is breastfeeding or pregnant.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) wine, 12 ounces (360 mL) of beer, or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening as disclosed by subject during evaluation

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects, aged 12-75 years old, with active mild to severe atopic dermatitis (AD)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Scratch Movements | 5 days
  To evaluate the agreement between the outcomes acquired by video annotation and accelerometry regarding scratch movement.
Sleep Time | 5 days
  To evaluate the agreement between the outcomes of amount of time asleep acquired by polysomnography, sleep sensor pad, and accelerometry.

SECONDARY OUTCOMES:
Sleep Efficiency | 5 days
  To evaluate the agreement between the outcomes of sleep efficiency acquired by polysomnography, sleep sensor pad and accelerometry.
Patient-Reported Outcomes/ Scratch | 5 days
  To evaluate the agreement between the scratch outcomes acquired by accelerometry and patient-reported outcome (PRO) measures (as measured by the scales of the respective PROs).
Patient-Reported Outcomes/ Sleep | 5 days
  To evaluate the agreement between the sleep outcomes acquired by accelerometry and patient-reported outcome (PRO) measures (as measured by the scales of the respective PROs).
Quality of Life/ Scratch | 5 days
  To evaluate the agreement between the scratch outcomes acquired by accelerometry and quality of life measures, as measured by scores of the Quality of Life Questionnaires.
Quality of Life/ Sleep | 5 days
  To evaluate the agreement between the sleep outcomes acquired by accelerometry and quality of life measures, as measured by scores of the Quality of Life Questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Beck, MD, Principal Investigator — University of Rochester; Earl R. Dorsey, MD MBA, Study Chair — University of Rochester Medical Center/Center for Health+Technology
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided